CLINICAL TRIAL: NCT03971617
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Safety and Tolerability of Molecular Hydrogen in Patients With Parkinson's Disease
Brief Title: Clinical Trial to Evaluate the Safety and Tolerability of Hydrogen in Patients With Parkinson's Disease
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Insufficient enrollment to answer research question
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Carine Maurer, Assistant Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H2PD
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Results first posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Hydrogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hydrogen tablets (Experimental): The ingredient in the tablet producing H2 is magnesium. Each tablet contains 80 mg magnesium, a safe level well below the recommended daily dietary allowance of 420 mg for men/ 320 mg for women. Dissolving one tablet in 250 mL of water will achieve a saturating H2 concentration of approximately 1.6 ppm. Twice a day subjects will dissolve a tablet into water and drink the effervescent water.
  Interventions: Drug: Hydrogen
- Placebo tablets (Placebo Comparator): effervescent placebo tablets will also contain 80 mg magnesium but do not generate hydrogen-enriched water
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Hydrogen — each hydrogen tablet contains 80mg magnesium
  Arms: Hydrogen tablets
Drug: Placebo oral tablet — matching placebo tablet
  Arms: Placebo tablets

SUMMARY:
This study is a placebo-controlled, double-blind trial that will investigate the safety and tolerability of molecular hydrogen, a promising antioxidant agent, in patients with early-stage Parkinson's Disease. The medication will be administered orally as 8 ounces of hydrogen-enriched drinking water twice a day over the course of one year.

DETAILED DESCRIPTION:
This study will investigate the safety and tolerability of molecular hydrogen, a promising antioxidant agent, in patients with early-stage Parkinson's Disease. Subjects will be sequentially randomized in a 1:1 ratio to receive hydrogen-enriched water or the corresponding placebo twice a day, in addition to all standard-of-care treatments. Enrollment goal is 70 subjects. Duration of therapy is 52 weeks.

The primary outcome measures are safety and tolerability of hydrogen-enriched water. Secondary outcome measures include: progression of motor symptoms, health-related quality of life, progression of cognitive decline, and progression of symptom burden.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease
* Modified Hoehn & Yahr Stage < III
* Diagnosis of Parkinson's Disease made within past 3 years•
* Ability to complete questionnaires
* Willingness to go off parkinsonian medication for 12 hours prior to baseline and 56-week assessments

Exclusion Criteria:

* Other major diseases of the central nervous system
* History of stroke
* Use of antipsychotic neuroleptic medication within the last 6 months
* Symptomatic (secondary) parkinsonism
* Atypical parkinsonian variants
* Unstable medical or psychiatric illness
* Known kidney disease
* History of stereotactic brain surgery
* Significant cognitive impairment
* Inability to safely tolerate 8 ounces of water twice daily associated with the study medication
* Unable to avoid regular use of medications containing magnesium
* Treatment with another investigational drug within the last 30 days that may interfere with the study medication
* Pregnancy or nursing

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carine Maurer, MD,PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Medical Center, Stony Brook, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydrogen Tablets | Placebo Tablets
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrogen Tablets | Placebo Tablets | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-emergent Adverse Events
Description: Number of treatment-emergent adverse events [safety and tolerability] of H2-enriched water in patients with Parkinson's disease (PD).
Time Frame: 56 weeks
Measure: Number; unit: Adverse Events
Arm/Group | Hydrogen Tablets | Placebo Tablets
Number analyzed (Participants) | 1 | 1
Adverse Events | 0 | 0

2. Secondary Outcome: Score on the Part III Subscale of the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
Description: Change from baseline to week 56 in motor examination, as assessed by score on Part III of the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS). Part III of the MDS-UPDRS assesses the motor signs of Parkinson's Disease. Scores range from 0-33 with a lower score indicating less severe impairment.
Time Frame: 56 weeks
Population: Note: Data cannot be reported due to privacy issues associated with low enrollment
Arm/Group | Hydrogen Tablets | Placebo Tablets
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Score on the Parkinson's Disease Quality of Life Questionnaire (PDQ-39)
Description: Change from baseline to week 56 in Parkinson's Disease-related quality of life as assessed by the Parkinson's Disease Quality of Life Questionnaire (PDQ-39). The PDQ-39 assesses how often patients experience difficulties across 8 quality of life domains (mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communication, and bodily discomfort). Scores for each domain range from 0 to 100 with lower scores indicating more impaired quality of life. The overall score is an average of the scores for the 8 dimensions.
Time Frame: 56 weeks
Population: Note: results cannot be reported due to privacy issues associated with low enrollment
Arm/Group | Hydrogen Tablets | Placebo Tablets
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Score on the Montreal Cognitive Assessment (MoCA)
Description: Change from baseline to week 56 in overall cognitive function as assessed by the Montreal Cognitive Assessment (MoCA) score. Scores on the MoCA range from 0-30 with lower scores indicating more cognitive impairment.
Time Frame: 56 weeks
Population: Note: Data cannot be reported due to privacy issues associated with low enrollment
Arm/Group | Hydrogen Tablets | Placebo Tablets
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Score on the Combined Part I, Part II, Part III, and Part IV Subscales of the Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
Description: Change from baseline to week 56 on the Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS). The MDS-UPDRS consists of four sub-scales. For each sub-scale, lower scores indicate less severe impairment. The scales are: Part I, non-motor experiences of daily living (scores range from 0-52); Part II, motor experiences of daily living (scores range from 0-52); Part III, motor examination (scores range from 0-132) and part IV, motor complications (scores range from 0-24). Score for the total assessment ranges from 0 to 260 with lower scores indicating less severe impairment.
Time Frame: 56 weeks
Population: Note: Data cannot be reported due to privacy issues associated with low enrollment
Arm/Group | Hydrogen Tablets | Placebo Tablets
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 56 Weeks
Arm/Group | Hydrogen Tablets | Placebo Tablets
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Due to low enrollment in this study, we are not able to report on study outcome measures for participants and are unable to draw conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT03971617/Prot_SAP_000.pdf